## MEASUREMENT FLOWCHART

Apply to the Sleep Disorders Centre for a sleep record.



The participant is invited to join the study.



Ţ

Participation in the study has been accepted.

Declined participation in the study.



Single-night measurement.

In addition to polysomnography (PSG),

- >A device combining EEG and PPG sensors is placed on the forehead.
  > PPG sensor placed on the wrist.



Data analysis:

- > Classification of PSG records by human experts.
- > Classification of the data from our sleep device with the classifier we have developed.



Comparison of Two Results:

- >Cohen's Kappa
- > F score calculation
- > Bland-Altman plots

We have 305 nights of sleep data from different individuals who may have possible sleep disorders. The dataset is described in Figure 1.

## **OUR DATASET**



Figure 1: A description of our datasets.